CLINICAL TRIAL: NCT00423436
Title: Using an Interactive Voice Response Telephone System in the Assessment and Management of Symptoms in Advanced Lung Cancer Patients Receiving Chemotherapy
Brief Title: Interactive Voice Response (IVR) Symptom Assessment in Non-Small Cell Lung Cancer (NSCLC) Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: ID01-243
Record Dates: First submitted 2007-01-16; First posted 2007-01-18 (Estimated); Results first posted 2011-12-16 (Estimated); Last update posted 2011-12-16 (Estimated); Status verified 2011-11

CONDITIONS: Lung Cancer
Keywords: Non-Small Cell Lung Cancer; Small Cell Lung Cancer; Voice Response System; Questionnaire; Survey; NSCLC
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung; Small Cell Lung Carcinoma | interventions — Surveys and Questionnaires; Triage

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- IVR Assessment Plus Triage (Experimental): Interactive Voice Response Telephone System (IVR) Plus Triage (Participants report symptoms to telephone system and doctor/nurse notified when symptom is severe) + Questionnaire
  Interventions: Behavioral: Questionnaire; Behavioral: Interactive Voice Response Telephone System; Behavioral: IVR Plus Triage
- IVR Assessment Only (Experimental): IVR (Phone calls twice weekly) + Questionnaire
  Interventions: Behavioral: Questionnaire

INTERVENTIONS:
Behavioral: Questionnaire — Questionnaires taking about 30-45 minutes to complete.
  Other Names: Survey
Behavioral: Interactive Voice Response Telephone System — IVR Only = Phone calls twice weekly, each call lasting less than 5 minutes.
  Arms: IVR Assessment Plus Triage
Behavioral: IVR Plus Triage — IVR system will "triage," or sort, the symptom data by symptom severity, notifying health care professionals when a symptom is greater than the set threshold limit.
  Other Names: interactive voice recognition; IVR
  Arms: IVR Assessment Plus Triage

SUMMARY:
Primary Objectives:

* To compare the effectiveness of an interactive voice response (IVR) telephone triage/feedback system versus an interactive voice response telephone system with assessment only in monitoring and managing symptoms in patients with advanced non small cell lung cancer (NSCLC).
* To compare differences in mood and quality of life variables of patients using the IVR triage/feedback system versus IVR assessment only.
* To compare the healthcare utilization (emergency visits, admissions, length of stay for hospitalizations for uncontrolled symptoms) of patients using the IVR triage/feedback system versus IVR assessment only.

DETAILED DESCRIPTION:
You will be asked to complete several questionnaires during a visit to the Thoracic Clinic. These questionnaires measure physical and emotional symptoms, and quality of life. Completing the questionnaires takes about 30-45 minutes. The research nurse will also teach you how to use the telephone system for reporting symptoms. You will tell the research nurse when the most convenient times for the telephone calls and the telephone system will be set up to call at those times.

It is not clear at this time whether the telephone symptom evaluation is better than the usual plan that doctors and nurses follow for asking about symptoms. For this reason, you will be randomly picked (as in the toss of a coin) to be in one of two groups. The chance of being in either one of the two programs is about equal.

Half of the patients will be assigned to the "telephone assessment system plus triage" group. If you are assigned to this group, you will report symptoms to the telephone system and the doctor or nurse at M.D. Anderson will be notified when a symptom is severe. You will also be encouraged to report all symptoms to their doctor and nurse at M.D. Anderson.

Half of the patients will be assigned to the "telephone assessment only" group. If you are assigned to this group, your symptom information will only be given through the telephone system. You will also be encouraged to report all symptoms directly to your doctor and nurse at M.D. Anderson. Your physician may request information from the telephone system.

If you are assigned to this "telephone assessment only" group, the telephone system will call you twice a week during 2 cycles of chemotherapy. It is programmed to ask you to rate your symptoms and how much the symptoms interfere in your life. Rating symptoms using the telephone system takes less than five minutes for each call.

After each chemotherapy cycle, you and patients in both groups will be asked to fill out questionnaires during a clinic visit. The questionnaires are used to measure emotional symptoms and quality of life. Completing the questionnaires takes about 15-30 minutes. Your medical charts will also be reviewed and information collected about medical history.

If you have agreed to participate in the companion caregiver study, the study staff will use your demographic and clinical data to study the influence of your symptoms on your caregiver's physical and mental health.

This is an investigational study. About 100 will be enrolled at M.D. Anderson Cancer Center. A total of 136 patients will take part in this multicenter study.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with stage III or IV non-small cell lung cancer (NSCLC) or small cell lung cancer (SCLC) (Patients who have received other prior chemotherapy are eligible.)
* 18 years of age or older
* English-speaking
* Lives in the United States
* Adequate vision and hearing to use the Interactive Voice Response (IVR) system
* Provides written informed consent

Exclusion Criteria:

* Current diagnosis of psychosis or dementia
* Patients unable to complete the assessment measures or unable to understand the purpose of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2003-04; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Charles Cleeland, PhD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- UT MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: 04/30/03 to 12/10/08. All participants recruited at UT MD Anderson Cancer Center.
Pre-assignment Details: Of 84 enrolled, 16 participants dropped out before baseline assessment, prior to group assignment. Baseline data analysis was done on the remaining 68 patients (35 in the intervention and 33 in the control group).
Period: Overall Study
Arm/Group | IVR Assessment Plus Triage | IVR Assessment Only
Started | 35 | 33
Completed | 35 | 33
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | IVR Assessment Plus Triage | IVR Assessment Only | Total
Number analyzed (Participants) | 35 | 33 | 68
Age Continuous [Mean (Standard Deviation); unit: years] | 64.41 (9.11) | 60.63 (8.40) | 62.5762 (8.9158)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 18 | 36
  Male | 17 | 15 | 32
Region of Enrollment [Number; unit: participants]
  United States | 35 | 33 | 68

OUTCOME MEASURES:

1. Primary Outcome: Ratio of Number of Alerts Generated by Symptom Distress Over the Number of Available Assessments
Description: Total number of alerts generated by symptom exceeding prespecified threshold for 7 symptoms - pain, fatigue, nausea, cough, constipation, vomiting and shortness of breath (Ratio alerts/number of assessments using IVR telephone triage/feedback versus IVR only). Reporting 0-10 severity scale of MD Anderson Symptom Inventory from 0 (symptom not present) to 10 (symptom bad as imagine it could be). Thresholds set at 4 on scale for all symptoms except shortness of breath and constipation where threshold set at 2. More than one symptom alert may appear per assessment causing ratio values to exceed 1.
Time Frame: Baseline to end of first chemotherapy cycle (generally chemotherapy and 1 assessment of response within 6-8 weeks)
Population: Analysis was per protocol. Due to attrition, data from 61 participants were analyzed at end of first chemotherapy cycle and from 27 participants at the end of the study.
Measure: Number; unit: Ratio of alerts/number of assessments
Units Other Than Participants: Alerts
Arm/Group | IVR Assessment Plus Triage | IVR Assessment Only
Number analyzed (Participants) | 35 | 33
Number analyzed (Alerts) | 100 | 200
Ratio of alerts/number of assessments | 0.96 | 1.56

ADVERSE EVENTS:
Time Frame: 5 years
Arm/Group | IVR Assessment Plus Triage | IVR Assessment Only
Serious Adverse Events (participants affected / at risk) | 0/35 | 0/33
Other Adverse Events (participants affected / at risk) | 0/35 | 0/33

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No